CLINICAL TRIAL: NCT02072356
Title: A Humanitarian Device Exemption Treatment Protocol of TheraSphere® For Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: Radiolabeled Glass Beads in Treating Patients With Liver Cancer That Cannot be Removed by Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Ali Rikabi, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-10036; NCI-2012-00877 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
Keywords: Humanitarian Device; Carcinoma; Hepatocellular Carcinoma; TheraSphere®; HUD
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment (yttrium Y 90 glass microspheres) (Experimental): Patients receive yttrium Y 90 glass microspheres IA on day 0. Patients may receive additional treatment 4-12 weeks after initial treatment at the discretion of the study physician.
  Interventions: Radiation: yttrium Y 90 glass microspheres; Other: laboratory biomarker analysis; Drug: TheraSphere

INTERVENTIONS:
Radiation: yttrium Y 90 glass microspheres — Given Interartrial
  Other Names: TheraSphere
Other: laboratory biomarker analysis — Alpha-fetoprotein assay
  Other Names: Correlative studies; AFP
Drug: TheraSphere — TheraSphere is delivered into the liver tumor through a catheter placed into the hepatic artery.

SUMMARY:
This clinical trial studies radiolabeled glass beads (yttrium Y 90 glass microspheres) in treating patients with unresectable hepatocellular carcinoma. Internal radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells. Using radiolabeled glass beads to kill tumor cells may be an effective treatment for liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Provide oversight to treatment with TheraSphere to eligible patients with hepatocellular carcinoma (HCC) of the liver who are not surgical resection candidates.

II. Evaluate patient experience, toxicities and overall survival associated with TheraSphere treatment.

OUTLINE:

Patients receive yttrium Y 90 glass microspheres intra-arterially (IA) on day 0, and may receive a second dose within 30-90 days of initial treatment. Patients may receive additional treatment 4-12 weeks after initial treatment at the discretion of the study physician.

After completion of study treatment, patients are followed up at 3-6 weeks and annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intrahepatic malignancy including but not limited to HCC; the histopathology confirmation criterion may be waived in patients with a radiographically identifiable liver mass, known laboratory or clinical risk factors for cancer or elevated tumor markers such as alpha-fetoprotein (AFP) and clinical findings
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 - 2
* Life expectancy >= 3 months
* > 4 weeks since prior radiation, surgery or chemotherapy
* Able to comprehend and provide written informed consent in accordance with institutional and federal guidelines
* Ineligible for surgical resection

Exclusion Criteria:

* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times upper limit of normal (UNL)
* Serum bilirubin > 2.0 mg/dl (unless segmental infusion is planned)
* Any contraindications to angiography and hepatic artery catheterization such as:

  * History of severe allergy or intolerance to any contrast media, narcotics, sedatives, or atropine that cannot be corrected or premedicated
  * Bleeding diathesis, not correctable by usual forms of therapy
  * Severe peripheral vascular disease that would preclude catheterization
* Evidence of potential delivery of greater than 16.5 mCi (30 Gy absorbed dose) of radiation to the lungs in a single treatment
* Evidence of pulmonary insufficiency
* Evidence of any detectable technetium-99m macroaggregated serum albumin (Tc-99m MAA) flow to the stomach or duodenum, not correctable by using established angiographic techniques to stop or mitigate such flow
* Significant extrahepatic disease representing an imminent life-threatening outcome
* Active uncontrolled infection
* Significant underlying medical or psychiatric illness
* Co-morbid disease of condition that would preclude safe delivery of TheraSphere treatment or, in the judgment of the physician, place the patient at undue risk
* Pregnancy

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2010-10-11 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Response to treatment | Up to 2 years
Survival time | Up to 2 years
Adverse experiences | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rikabi Ali, M.D., Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu